CLINICAL TRIAL: NCT05667324
Title: Post-operative Pain Control With Sphenopalantine Ganglion Nerve Block in Septorhinoplasty Patients
Brief Title: Septorhinoplasty Post-operative Pain Control With SPG Nerve Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202201279 -A
Record Dates: First submitted 2022-11-04; First posted 2022-12-28 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Deviated Nasal Septum
Keywords: Post-op pain; septorhinoplasty; deviated septum
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Ropivacaine plus Dexamethasone (Experimental): The group 1 injection procedure will be performed as follows: after preparation of the skin using appropriate skin preparation solution and using aseptic technique, a small-gauge spinal needle will be advanced into the pterygopalatine fossa under ultrasound guidance. Once the needle is properly positioned, 0.5% ropivacaine will be administered at a dose of 20 mg plus 4 mg dexamethasone and the needle will be removed. This procedure will be performed bilaterally
  Interventions: Drug: Ropivacaine; Drug: Dexamethasone
- Group 2: Placebo plus Dexamethasone (Active Comparator): In group 2 the same procedure will be performed, but the injectate will consist of 5 mL of a balanced crystalloid intravenous solution (4 ml of normal saline) plus 4 mg dexamethasone (each side). This procedure will be performed bilaterally.
  Interventions: Drug: Dexamethasone; Drug: Placebo

INTERVENTIONS:
Drug: Ropivacaine — A single injection into the pterygopalatine fossa bilaterally of 0.5% ropivacaine at a dose of 20 mg (each side)
  Arms: Group 1: Ropivacaine plus Dexamethasone
Drug: Dexamethasone — Plus 4 mg dexamethasone
Drug: Placebo — A single injection into the pterygopalatine fossa bilaterally of a balanced crystalloid intravenous solution (4 ml of normal saline)
  Arms: Group 2: Placebo plus Dexamethasone

SUMMARY:
Maxillary nerve blocks have been shown to significantly reduce post-operative pain and analgesic intake during the 24-hour period following sinus surgery. This randomized, double-blinded, placebo-controlled study will investigate blocks of the pterygopalatine fossa using a suprazygomatic approach during septorhinoplasty surgery. It is the investigator's hypothesis that this technique will result in decreased post-operative pain and opioid use, and the morbidity associated with it.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting for open or endoscopic septorhinoplasty
* Age 18-80
* Normal oral food and water intake before surgery
* ASA physical classification 1-3

Exclusion Criteria:

* Refusal to consent
* Patients without a cellular phone or who are unable to accept text messages
* Allergy to opioid narcotics
* ASA physical classification of 4 or higher
* Patient requires other surgery in addition to septorhinoplasty
* Age > 80 or <18
* Any underlying chronic pain condition or ongoing opioid use over the preceding 3 months
* Presence of any other factor which, at the discretion of any member of the study team, makes the patient a poor candidate for block placement.
* Presence of any other factor which, at the discretion of any member of the study team, makes the patient a poor candidate for research participation.
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Decrease the opioid requirement post-operatively as assessed by providers. | 7 days +/- 2 days
  post operative period

SECONDARY OUTCOMES:
Decrease in post-anesthesia care unit observation time. | 60-180 minutes
  PACU duration times
Efficiency of SMS based survey for post-operative data collection. | 5 days post-operatively +/- 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Johnson, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health of University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No